CLINICAL TRIAL: NCT01685931
Title: Effectiveness, Safety and Tolerability of Flexibly Dosed Paliperidone Palmitate in Patients With Schizophrenia Previously Unsuccessfully Treated by Oral Antipsychotics and With Acute Symptom of Schizophrenia: A 13-Week, Open-label, Single-arm, Multicenter, Prospective, Interventional Study Followed by a Naturalistic Additional 1 Year Follow up
Brief Title: A Study of Paliperidone Palmitate in Patients With Schizophrenia Previously Unsuccessfully Treated by Oral Antipsychotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100880; R092670SCH4019 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2012-09-11; First posted 2012-09-14 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Palmitate; Oral Antipsychotics; Invega Sustenna
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone Palmitate (Experimental)
  Interventions: Drug: Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone Palmitate — One intramuscular injection of paliperidone palmitate flexible dose will be administered on Day 1, Day 8, and monthly thereafter.

SUMMARY:
The purpose of this study is to assess the effectiveness, safety and tolerability of flexibly dosed paliperidone palmitate in patients with schizophrenia previously unsuccessfully treated by oral antipsychotics and with acute symptom of schizophrenia.

DETAILED DESCRIPTION:
This is a 13-week, open-label (all people know the identity of the intervention), single-arm (one group of patients), multicenter, prospective, interventional study in Chinese patients. In a prospective, interventional study, the patients identified receive a treatment during the course of the research study and are followed forward in time for the outcome of the study. In China, there is still insufficient information about effectiveness, tolerability, and dosage strategy for directly switching from previous oral antipsychotics (drugs that are helpful in the treatment of psychosis and have a capacity to ameliorate thought disorders) in patients with acute symptoms. Acute symptoms are quick and severe form of illness in its early stage. In addition, there is also lack of information about bridging acute phase to long-term treatment. In this study, patients with multiple types of acute schizophrenia will be recruited and will receive Sustenna (paliperidone palmitate) treatments for 13 weeks. After the acute treatment, the patients will continue to receive the prescribed medication and will be followed up for an additional 52 weeks to assess the outcomes related to long-term treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of schizophrenia
* Experiencing an acute episode, with a Positive and Negative Syndrome Scale (PANSS) total score between 70 and 120, inclusive
* Patients currently treated with antipsychotic are allowed to be recruited
* Be medically stable on the basis of clinical laboratory tests performed at screening

Exclusion Criteria:

* A primary diagnosis other than schizophrenia
* History of risperidone or paliperidone resistance as defined by failure to respond to 2 adequate treatment periods
* Clozapine use for treatment refractory schizophrenia
* Relevant history or current presence of any significant or unstable condition, disease or illness that could limit the participation in the study according to the investigator
* Woman who is pregnant, breast-feeding, or is planning to become pregnant within 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with a 30% reduction from baseline in Positive and Negative Syndrome Scale (PANSS) | Baseline, Week 13
  The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.

SECONDARY OUTCOMES:
The change from baseline in Positive and Negative Syndrome Scale (PANSS) score | Baseline, Week 13
  The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.
The change from baseline in Clinical Global Impression - Severity (CGI-S) | Baseline, Week 13
  The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill patients". Higher scores indicate worsening.
The change from baseline in Medication Satisfaction Questionnaire (MSQ) | Baseline, Week 13
  The MSQ is a 7-point, Likert-type scale rated as follows: 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Somewhat Dissatisfied, 4=Neither Satisfied or Dissatisfied, 5=Somewhat Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. Worst value is 1 (Extremely Dissatisfied) and best value is 7 (Extremely Satisfied).
The change from baseline in Involvement Evaluation Questionnaire (IEQ) | Baseline, Week 13
  The IEQ is a 31-item questionnaire that assesses the encouragement and care that the caregiver has to give to the patient, to personal problems between patient and caregiver, and to the caregiver's worries, coping and subjective burden. All items are scored on 5-point Likert scales (never, sometimes, regularly, often, always).
The change from baseline in Medication Adherence Rating Scale (MARS) | Baseline, Week 13
  The MARS is a ten-item yes/no self-report measure of medication adherence in psychosis. Total scores range from 0 (low likelihood of medication adherence) to 10 (high likelihood of medication adherence).
The change from baseline in Medication Preference Questionnaire (MPQ) | Baseline, Week 13
  The MPQ is used to investigate which treatment (oral or injection) the patients prefer and why they prefer this treatment, and to investigate which injectable site (deltoid or gluteal) they prefer and why they prefer this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (17):
- China (17):
  - Baoding
  - Beijing
  - Chengdu
  - Chongqing
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Jinan
  - Nanjing
  - Qingdao
  - Shantou
  - Shenzhen
  - Shijiazhuang
  - Suzhou
  - Taiyuan
  - Tianjin
  - Wuhan

REFERENCES:
- See also: A Study of Paliperidone Palmitate in Patients with Schizophrenia Previously Unsuccessfully Treated by Oral Antipsychotics — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3548&filename=CR100880_CSR.pdf